CLINICAL TRIAL: NCT00466193
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study of the Efficacy and Safety of the Zolpidem Tartrate Sublingual Tablet in Adult Subjects With Insomnia Characterized by Difficulty Returning to Sleep After Awakening in the Middle-of-the-Night (MOTN)
Brief Title: A Study of Zolpidem Tartrate Sublingual Tablet in Adult Patients With Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Transcept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZI-12
Record Dates: First submitted 2007-04-24; First posted 2007-04-27 (Estimated); Results first posted 2012-01-20 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Insomnia
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zolpidem 3.5mg (Experimental)
  Interventions: Drug: zolpidem tartrate sublingual tablet
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: zolpidem tartrate sublingual tablet — 3.5 milligram zolpidem tartrate sublingual tablet taken as needed following a middle-of-the-night awakening over the 28-night study period. Participants placed the study drug under the tongue and allowed it to dissolve there for about 2 minutes, then swallowed after dissolved.
  Other Names: Intermezzo®
  Arms: Zolpidem 3.5mg
Drug: Placebo — Placebo sublingual tablet taken as needed following a middle-of-the-night awakening over the 28-night study period. Participants placed the study drug under the tongue and allowed it to dissolve there for about 2 minutes, then swallowed after dissolved.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate sleep onset following administration of zolpidem tartrate sublingual tablet (Intermezzo) versus placebo in adult insomnia patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults with history of sleeplessness

Exclusion Criteria:

* Allergic to investigational drug
* Any conditions and medications that may interfere with study drug evaluation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 295 (Actual)
Dates: Start 2007-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krystal, MD, Principal Investigator — Clinical Neurophysiology Training Program, Duke University; Thomas Roth, PhD, Principal Investigator — Sleep Disorders and Research Center, Henry Ford Hospital
Locations (1):
- Transcept Investigational Site, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seven hundred and three (703) subjects were screened. Three hundred (300) subjects were randomized, but 5 subjects never took drug.
Groups:
- Zolpidem 3.5 mg: Zolpidem tartrate sublingual tablet, 3.5 milligram, taken following a middle-of-the-night awakening.
- Placebo: Placebo sublingual tablet taken following a middle-of-the-night awakening.
Period: Overall Study
Arm/Group | Zolpidem 3.5 mg | Placebo
Started | 150 | 145
Completed | 138 | 137 (One patient did not report at least one Latency Sleep Onset following middle-of-the-night awakening.)
Not Completed | 12 | 8
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Patient refused Visit 4 procedures | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zolpidem 3.5 mg | Placebo | Total
Number analyzed (Participants) | 150 | 145 | 295
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 150 | 145 | 295
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.3 (11.38) | 43.4 (11.30) | 42.8 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 94 | 201
  Male | 43 | 51 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 47 | 45 | 92
  White | 96 | 94 | 190
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 150 | 145 | 295
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilogram per square meter | 26.17 (3.860) | 26.55 (3.754) | 26.35 (3.807)
Weight [Mean (Standard Deviation); unit: kilograms] | 74.27 (15.050) | 75.73 (13.434) | 74.99 (14.273)

OUTCOME MEASURES:

1. Primary Outcome: Latency to Sleep Onset After Middle-of-the-Night Awakening at Baseline
Description: Time was recorded by study participants using a telephone interactive voice response system (IVRS) to answer the question: How long did it take you to fall asleep after taking your study medication?
Time Frame: Weeks -1 to 0
Population: Efficacy population: randomized participants who took at least one dose of study medication and had at least one latency to sleep onset following a middle-of-the-night awakening value.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem 3.5 mg | Placebo
Number analyzed (Participants) | 150 | 144
minutes | 68.13 [63.90 to 72.64] | 69.42 [65.03 to 74.10]

2. Secondary Outcome: Subjective Total Sleep Time Following Middle-of-the-Night Awakening at Baseline
Description: Total sleep time in minutes after waking in the middle of the night. The values were recorded by participants using a telephone interactive voice response system (IVRS) to answer the question: After you fell back to sleep, how long did you sleep until you woke up this morning?
Time Frame: Weeks -1 to 0
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem 3.5 mg | Placebo
Number analyzed (Participants) | 150 | 144
minutes | 241.2 [229.1 to 253.4] | 222.9 [210.5 to 235.3]

3. Secondary Outcome: Subjective Total Sleep Time Following Middle-of-the-Night Awakening During Double-blind Treatment
Description: as for outcome 2
Time Frame: Weeks 1 to 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem 3.5 mg | Placebo
Number analyzed (Participants) | 150 | 144
minutes | 264.1 [255.7 to 272.4] | 255.0 [246.5 to 263.5]

4. Secondary Outcome: Subjective Number of Awakenings Following Middle-of-the-Night Awakening at Baseline.
Description: Number of awakenings following middle-of-the-night awakening were recorded by study participants using a telephone interactive voice response system (IVRS) to answer the question: After you fell back to sleep, how many times did you wake up again before waking up in the morning?
Time Frame: Weeks -1 to 0
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Zolpidem 3.5 mg | Placebo
Number analyzed (Participants) | 150 | 144
percentage of participants
  0 awakenings | 16.7 | 11.8
  >0 and <=1 awakenings | 46.0 | 45.1
  >1 and <=2 awakenings | 26.0 | 27.1
  >2 awakenings | 11.3 | 16.0

5. Secondary Outcome: Subjective Number of Awakenings Following Middle-of-the-Night Awakening During Double-blind Treatment
Description: as for outcome 4
Time Frame: Weeks 1 to 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Zolpidem 3.5 mg | Placebo
Number analyzed (Participants) | 150 | 144
percentage of participants
  0 awakenings | 30.0 | 16.7
  >0 and <=1 awakenings | 46.0 | 43.1
  >1 and <=2 awakenings | 17.3 | 25.0
  >2 awakenings | 6.7 | 15.3
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for treatment

6. Secondary Outcome: Subjective Wake Time After Sleep Onset Following Middle-of-the-Night Awakening at Baseline
Description: The number of minutes subjects reported being awake after onset of sleep following middle-of-the-night awakening during the baseline period. Values were recorded using a telephone interactive voice response system (IVRS) to answer the question: Considering all of these awakenings (after taking study medication and returning to sleep), how long were you awake from the time you went back to sleep after dosing until you got out of bed this morning?
Time Frame: Weeks -1 to 0
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Zolpidem 3.5 mg | Placebo
Number analyzed (Participants) | 150 | 144
percentage of participants
  No wake time | 16.7 | 11.8
  >0 to 20 minutes | 18.7 | 14.6
  21 to 60 minutes | 25.3 | 32.6
  >60 minutes | 39.3 | 41.0

7. Secondary Outcome: Subjective Wake Time After Sleep Onset Following Middle-of-the-Night Awakening During Double-blind Treatment
Description: The number of minutes subjects reported being awake after onset of sleep following middle-of-the-night awakening during double-blind treatment. Values were recorded using a telephone interactive voice response system (IVRS) to answer the question: Considering all of these awakenings (after taking study medication and returning to sleep), how long were you awake from the time you went back to sleep after dosing until you got out of bed this morning?
Time Frame: Weeks 1 to 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Zolpidem 3.5 mg | Placebo
Number analyzed (Participants) | 150 | 144
percentage of participants
  No wake time | 30.0 | 16.7
  >0 to 20 minutes | 27.3 | 26.4
  21 to 60 minutes | 26.0 | 31.9
  > 60 minutes | 16.7 | 25.0
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Placebo; Test type: Superiority or Other; p = 0.006, ANCOVA — p-value is for treatment

8. Secondary Outcome: Morning Sleepiness Rating Following Dosing Post Middle-of-the-Night Awakening at Baseline
Description: Morning sleepiness was assessed using a 9-point sleepiness scale (1=very sleepy to 9=wide awake and alert). During the baseline period, all participants received placebo.
Time Frame: Weeks -1 to 0
Population: Safety population: participants who took at least one dose of study medication post-randomization.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Zolpidem 3.5 mg | Placebo
Number analyzed (Participants) | 150 | 145
units on a scale | 4.87 [4.61 to 5.13] | 4.71 [4.45 to 4.97]

9. Primary Outcome: Latency to Sleep Onset After Middle-of-the-Night Awakening During Double-blind Treatment
Description: as for outcome 1
Time Frame: Weeks 1 to 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem 3.5 mg | Placebo
Number analyzed (Participants) | 150 | 144
minutes | 38.22 [35.06 to 41.66] | 56.37 [51.63 to 61.56]

10. Secondary Outcome: Morning Sleepiness Rating Following Dosing Post Middle-of-the-Night Awakening During Double-blind Treatment
Description: Morning sleepiness was assessed using a 9-point sleepiness scale (1=very sleepy to 9=wide awake and alert). Values are from dosing nights during double-blind treatment.
Time Frame: Weeks 1 to 4
Population: Safety population: participants who took at least one dose of study medication post-randomization.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Zolpidem 3.5 mg | Placebo
Number analyzed (Participants) | 150 | 145
units on a scale | 5.59 [5.42 to 5.76] | 5.24 [5.06 to 5.41]
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0041, ANCOVA — P-value is for treatment

ADVERSE EVENTS:
Time Frame: Weeks 1-4
Arm/Group | Zolpidem 3.5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/145
Other Adverse Events (participants affected / at risk) | 0/150 | 0/145

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor agrees to review manuscripts within sixty (60) days prior to submission for publication. If sponsor determines the publication includes patentable subject matter, sponsor may take an additional sixty (60) days to permit the filing of any patent applications.